CLINICAL TRIAL: NCT04543890
Title: A Multicenter, Prospective, Randomized Study Comparing Hypofractionated Radiotherapy With Hyperfractionated Radiotherapy Combined With Concurrent Chemotherapy and Omitting Clinical Target Volumes of the Primary Tumor in Limited-stage SCLC
Brief Title: A Prospective Study Comparing Two Radiotherapy Dose/Fraction and Omitting CTVs of the Primary Tumor in Limited SCLC
Acronym: CTV
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zhejiang Cancer Hospital (Other)
Collaborators: First Affiliated Hospital, Sun Yat-Sen University (Other); Chinese PLA General Hospital (Other); Guangdong Medical College (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB-2018-129
Record Dates: First submitted 2020-08-23; First posted 2020-09-10 (Actual); Last update posted 2020-09-10 (Actual); Status verified 2020-09

CONDITIONS: Small Cell Lung Cancer Limited Stage
Keywords: radiotherapy; chemotherapy; radiation dose; radiotherapy target volume
MeSH Terms: interventions — Radiation Dose Hypofractionation; Etoposide; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hyperfrationated Arm (Active Comparator): Patients with limited-stage SCLC receive etoposide and cisplatin (carboplatin) induction therapy for 2 cycles and then receive thoracic radiotherapy (45 Gy/30 fractions) with concurrent EP/EC chemotherapy for 2cycles, the CTVs of the tumor in lung parenchyma are omitted. Patients who achieve CR or PR then receive prophylactic cranial irradiation (PCI, 25 Gy/10 fractions).
  Interventions: Radiation: Hyperfractionated radiotherapy; Drug: Etoposide; Drug: Cisplatin
- Hypofrationated Arm (Experimental): Patients with limited-stage SCLC receive etoposide and cisplatin (carboplatin) induction therapy for 2 cycles and then receive thoracic radiotherapy (45 Gy/15 fractions) with concurrent EP/EC chemotherapy for 2cycles, the CTVs of the tumor in lung parenchyma are omitted. Patients who achieve CR or PR then receive prophylactic cranial irradiation (PCI, 25 Gy/10 fractions).
  Interventions: Radiation: Hypofractionated radiotherapy; Drug: Etoposide; Drug: Cisplatin

INTERVENTIONS:
Radiation: Hyperfractionated radiotherapy — Thoracic radiotherapy (45 Gy/30 fractions) for the Hyperfractionated Arm and prophylactic cranial irradiation (25 Gy/10 fractions).
  Arms: Hyperfrationated Arm
Radiation: Hypofractionated radiotherapy — Thoracic radiotherapy (45 Gy/15 fractions) for the Hypofractionated Arm and prophylactic cranial irradiation (25 Gy/10 fractions).
  Arms: Hypofrationated Arm
Drug: Etoposide — Etoposide will be administered IV 100mg/m2 on days 1-3, 22-24, 43-45 and 64-66.
  Other Names: VP-16
Drug: Cisplatin — Cisplatin will be administered IV 80mg/m2 on days 1, 22, 43 and 64.
  Other Names: DDP

SUMMARY:
For most of the patients with limited-stage SCLC, thoracic radiotherapy combined with chemotherapy is the standard treatment at present. However, the optimal dose / fraction of thoracic radiotherapy for limited-stage SCLC is still in controversial.This study is designed as a prospecitive randomized non-inferiority trial.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically/cytologically confirmed diagnosis of SCLC.
2. Radiologically (including brain CT/MRI, chest and abdomen contrasted CT and bone scintigraphy. PET/CT is recommended) confirmed limited-stage.
3. Patients should be between 18 and 75 years old.
4. ECOG performance status of 0-1 (Karnofsky performance status ≥ 80).
5. With adequate cardiac, pulmonary, bone marrow, hepatic and renal function.
6. With weight loss no more than 10% within 6 months before diagnosis.
7. Informed consent must be signed.

Exclusion Criteria:

1. Histology confirmed the mixed NSCLC components;
2. Other primary malignant tumors appeared within 5 years before the first administration of the study drug, except for locally curable malignant tumors after radical treatment (such as basal or squamous cell skin cancer, superficial bladder cancer or prostate, cervical or breast carcinoma in situ, etc.);
3. Any disease or condition contraindicated by radiotherapy or chemotherapy;
4. Malignant pleural effusion and pericardial effusion;
5. Pregnant and lactating women;
6. The investigator believes that the subject's complications or other circumstances may affect the compliance with the protocol or may not be suitable for the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2018-05-01 (Actual); Primary Completion 2023-06-01 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival | 2 years
  PFS, defined as the time from the date of randomization to the first date of documented objective progression disease or of death from any cause.

SECONDARY OUTCOMES:
Overall survival | 5 years
  OS, measured from the date of randomization to the date of death from any cause.

CONTACTS AND LOCATIONS:
Locations (1):
- Zhejiang Cancer Hospital, Hangzhou, Zhejiang, China